CLINICAL TRIAL: NCT02533453
Title: A 12/24-weeks, Open, Multi-centre, Phase IV Study on Safety and Efficacy of 2mg Exenatide Once Weekly (Bydureon) in Patients With Type 2 Diabetes Mellitus
Brief Title: A 12/24-weeks, Open, Multi-centre, Phase IV Study on Safety and Efficacy of 2mg Exenatide Once Weekly (Bydureon) in T2DM Patients.
Acronym: Bydureon
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5551L00018
Record Dates: First submitted 2015-08-11; First posted 2015-08-26 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus, T2DM, GLP-1, GLP-1 Once weekly, Exenatide
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bydureon (Experimental): exenatide once weekly
  Interventions: Biological: Bydureon

INTERVENTIONS:
Biological: Bydureon — exenatide once weekly
  Other Names: exenatide

SUMMARY:
As current study is conducted to provide additional information regarding safety and efficacy Bydureon, exenatide once weekly for injectable suspension, in the Korean population open label, non-comparative, multi-centre design is used.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 19-75 years of age
* diagnosed with type 2 diabetes mellitus
* Patients who have not achieved adequate glycaemic control on maximally tolerated doses of these oral therapies;

  * Metformin
  * Sulphonylurea
  * Thiazolidinedione
  * Metformin and sulphonylurea
  * Metformin and thiazolidinedione

Exclusion Criteria:

* Has been treated, is currently being treated, or is expected to require or undergo treatment with any of the following medications:

  1. Alpha glucosidase inhibitor or meglitinide within 30 days of screening;
  2. Insulin within 2 weeks prior to screening or insulin for longer than 1 week within 3 months of screening;
  3. DPP-4 inhibitors within 30 days of screening;
  4. Regular use (> 14 days) of drugs that directly affect gastrointestinal motility within 3 months of screening;
  5. Regular use (> 14 days) of systemic corticosteroids by oral, intravenous, or intramuscular route; or potent, inhaled, or intrapulmonary steroids known to have a high rate of systemic absorption within 3 months of screening;
  6. GLP-1 receptor agonist except exenatide within 3 months of screening;
* diagnosed with type 1 diabetes mellitus or diabetic ketoacidosis;
* type 2 diabetes by beta-cell dysfunction requiring insulin treatment
* Has ever used exenatide
* Pregnant or breast feeding patients
* Hepatic disease (defined by aspartate or alanine transaminase >3.0 times the upper limit of normal
* End-stage renal disease or severe renal impairment (creatinine clearance < 30 ml/min)

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-01-28 (Actual); Primary Completion 2016-12-07 (Actual); Study Completion 2016-12-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- South Korea (9):
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Gwangju
  - Research Site, Incheon
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Suwon
  - Research Site, Wŏnju

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from 15 hospitals in South Korea between Jan 2016 and Jul 2016.
Pre-assignment Details: 115 subjects were participated: 5 failed screening without treatment with the study drug.
Groups:
- 12/24 Weeks Treatment: Exenatide 2mg / 12/24 weeks treatment
Period: Overall Study
Arm/Group | 12/24 Weeks Treatment
Started | 110
Completed | 101
Not Completed | 9
Not completed — Adverse Event | 6
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: 104 were included in the safety set with 3 of inclusion/exclusion criteria deviations, 2 of treatment with prohibited concomitant medications, and 1 of enrolment before IRB approval excluded
Arm/Group | 12/24 Weeks Treatment
Number analyzed (Participants) | 104
Age, Customized [Count of Participants; unit: Participants]
  <50 years | 44
  Between 50 and 69 years | 58
  >=70 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 42

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events(AEs) and Serious Adverse Event(SAEs)
Description: was to estimate the incidence rates of adverse events (AEs) and serious adverse events (SAEs) in patients who are treated with 2 mg exenatide once weekly for type 2 diabetes mellitus in the normal clinical practice setting over a period of 12/24 weeks for long-term surveillance.
Time Frame: baseline and 12/24 weeks
Population: Of 110 subjects, 104 were included in the safety set with 3 of inclusion/exclusion criteria deviations, 2 of treatment with prohibited concomitant medications, and 1 of enrolment before IRB approval excluded.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 12/24 Weeks Treatment
Number analyzed (Participants) | 104
percentage of participants
  rate of all AEs | 52.9 [42.9 to 62.6]
  rate of all SAEs | 3.8 [1.04 to 9.38]

2. Secondary Outcome: Change in HbA1c
Description: Change in HbA1c at 12 and 24 weeks from start of the treatment(24 weeks just for patients allocated in long-term treatment)
Time Frame: baseline and 12/24 weeks
Population: Of 110 subjects, 104 were included in the safety set with 3 of inclusion/exclusion criteria deviations, 2 of treatment with prohibited concomitant medications, and 1 of enrolment before IRB approval excluded. Of 104 subjects, 1 subject who failed to receive the efficacy analysis was excluded, and 103 were included in the efficacy set.
Measure: Mean (Standard Deviation); unit: percentage of Hba1c
Arm/Group | 12/24 Weeks Treatment
Number analyzed (Participants) | 103
percentage of Hba1c | -1.21 (1.10)

3. Secondary Outcome: Change in Fasting Plasma Gloucose
Description: Change in Fasting plasma gloucose at 12 and 24 weeks from start of the treatment(24 weeks just for patients allocated in long-term treatment)
Time Frame: baseline and 12/24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 12/24 Weeks Treatment
Number analyzed (Participants) | 103
mg/dL | -34.2 (48.3)

4. Secondary Outcome: Change in Body Weight
Description: Change in body weight at 12 and 24 weeks from start of the treatment(24 weeks just for patients allocated in long-term treatment)
Time Frame: baseline and 12/24 weeks
Population: Of 110 subjects, 104 were included in the safety set with 5 subjects of non-treatment with the study drug, 3 of inclusion/exclusion criteria deviations, 2 of treatment with prohibited concomitant medications, and 1 of enrolment before IRB approval excluded.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | 12/24 Weeks Treatment
Number analyzed (Participants) | 104
kg | -0.95 (2.86)

5. Secondary Outcome: Change in Vital Sign
Description: Change in vital sign at 12 and 24 weeks from start of the treatment(24 weeks just for patients allocated in long-term treatment)
Time Frame: baseline and 12/24 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 12/24 Weeks Treatment
Number analyzed (Participants) | 104
mmHg
  SBP | -3.35 (11.95)
  DBP | -0.15 (9.58)

6. Secondary Outcome: Evaluation of "Subjective Improvement of Main Indication"
Description: "Subjective improvement of main indication" will be assessed as "improved," "slightly improved," "unchanged," "aggravated," or "unable to evaluate."
Time Frame: baseline and 12/24 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | 12/24 Weeks Treatment
Number analyzed (Participants) | 103
participants
  Improved | 84
  Slightly improved | 11
  Unchanged | 6
  Aggravated | 1
  unable to evaluate | 1

ADVERSE EVENTS:
Time Frame: 12 weeks / 24 weeks
Description: Of 110 subjects, 104 were included in the safety set with 3 of inclusion/exclusion criteria deviations, 2 of treatment with prohibited concomitant medications, and 1 of enrolment before IRB approval excluded.
Arm/Group | 12/24 Weeks Treatment
Serious Adverse Events (participants affected / at risk) | 4/104
Other Adverse Events (participants affected / at risk) | 55/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 12/24 Weeks Treatment (N=104)
Neuroendocrine tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Acute gastroenteritis (Infections and infestations) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 1 (1)
Hyperglycemia including diarrhea (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 12/24 Weeks Treatment (N=104)
Nausea (Gastrointestinal disorders) | 15 (16) — Of 110 subjects, 104 were included in the safety set with 3 of inclusion/exclusion criteria deviations, 2 of treatment with prohibited concomitant medications, and 1 of enrolment before IRB approval excluded.
Injection site nodule (General disorders) | 16 (16) — Of 110 subjects, 104 were included in the safety set with 3 of inclusion/exclusion criteria deviations, 2 of treatment with prohibited concomitant medications, and 1 of enrolment before IRB approval excluded.
Vomiting (Gastrointestinal disorders) | 9 (17) — Of 110 subjects, 104 were included in the safety set with 3 of inclusion/exclusion criteria deviations, 2 of treatment with prohibited concomitant medications, and 1 of enrolment before IRB approval excluded.
Diarrhoea (Gastrointestinal disorders) | 7 (11) — Of 110 subjects, 104 were included in the safety set with 3 of inclusion/exclusion criteria deviations, 2 of treatment with prohibited concomitant medications, and 1 of enrolment before IRB approval excluded.
injection site pruritus (General disorders) | 8 (8) — Of 110 subjects, 104 were included in the safety set with 3 of inclusion/exclusion criteria deviations, 2 of treatment with prohibited concomitant medications, and 1 of enrolment before IRB approval excluded.
Dizziness (Nervous system disorders) | 6 (10) — Of 110 subjects, 104 were included in the safety set with 3 of inclusion/exclusion criteria deviations, 2 of treatment with prohibited concomitant medications, and 1 of enrolment before IRB approval excluded.
Headache (Nervous system disorders) | 6 (10) — Of 110 subjects, 104 were included in the safety set with 3 of inclusion/exclusion criteria deviations, 2 of treatment with prohibited concomitant medications, and 1 of enrolment before IRB approval excluded.
Hypoglycaemia (Metabolism and nutrition disorders) | 7 (10) — Of 110 subjects, 104 were included in the safety set with 3 of inclusion/exclusion criteria deviations, 2 of treatment with prohibited concomitant medications, and 1 of enrolment before IRB approval excluded.
Decreased appetite (Metabolism and nutrition disorders) | 6 (8) — Of 110 subjects, 104 were included in the safety set with 3 of inclusion/exclusion criteria deviations, 2 of treatment with prohibited concomitant medications, and 1 of enrolment before IRB approval excluded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* The Institution and PI shall provide the Company with copies of any materials relating to the Study that either intends to publish (or submit for publication) or make any presentations relating to, at least 30 days in advance of publication
* At the request of the Company, the Institution and PI shall withhold publication for a period of 90 days from the date on which the Company receives the material.